CLINICAL TRIAL: NCT05661929
Title: The Association of Cognitive Distortions and NCDs Among Users of Medical Internet Resources
Status: Completed | Type: Observational
Sponsor: Limited Liability Company "Docstarclub" (Other)
Responsible Party: Sponsor
Other Study IDs: dsc001
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Cognitive Biases; Non-infecious Chronic Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Users of medical internet resources: This group includes people older 18 years who are looking for medical information at the Internet-resources
  Interventions: Other: Questionnaire CMQ

INTERVENTIONS:
Other: Questionnaire CMQ — The questionnaire is used to diagnose cognitive distortions. It includes 50 items to identify 10 the most common cognitive biases.

SUMMARY:
Currently, medical Internet resources are popular among the population of most countries, including Russia. So its can be used as a platform for mass measures of prevention.

Now we can receive a lot of information about socio-demographic characteristics, risk factors and the presence of chronic non-infectious diseases among users of medical Internet resources. And these knowledges are necessary to create effective online interventions for prevention of the most common diseases.

We have enough resources to identify and control risk factors for chronic non-infectious diseases. But adherence to doctor's recommendations remains at a low level. Working with cognitive biases is one of the points of application for increasing adherence to treatment and the rules of a healthy lifestyle.

Certain groups of patients have special cognitive biases. We assume that creation a typical portrait of a patient can reveal relationships and factors the variant of cognitive biases. This information may help to more effectively carry out preventive work with users of medical Internet resources, forming the correct patterns of perception and thereby improving adherence to the doctor's recommendations.

ELIGIBILITY:
Inclusion Criteria:

* User of medical Internet resources older 18 years

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: User of medical Internet resources
Sampling Method: Non-Probability Sample
Enrollment: 863 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
The questionnaire "Cognitive Mistakes Questionnaire" | from 1 February to 1 March 2022
  The questionnaire consist of 10 blocks on various types of cognitive distortions. Each block includes 5 questions. The maximum score of scale is 5 point, the minimum score of scale is 0 points. The maximum score means the severity of certain cognitive distortion

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Bezzubtseva, Study Director — Limited Liability Company "Docstarclub"
Locations (1):
- Limited Liability Company "Docstarclub", Sevastopol’, Russia